CLINICAL TRIAL: NCT01390337
Title: A Phase 1 Study of AC220 (ASP2689) in Combination With Induction and Consolidation Chemotherapy in Patients With Newly Diagnosed Acute Myeloid Leukemia
Brief Title: A Study to Assess AC220 Given in Combination With Induction and Consolidation Therapy in Newly Diagnosed Acute Myeloid Leukemia (AML)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Collaborators: Ambit Biosciences Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2689-CL-0005
Record Dates: First submitted 2011-07-07; First posted 2011-07-11 (Estimated); Last update posted 2019-02-12 (Actual); Status verified 2015-10

CONDITIONS: Leukemia, Myeloid, Acute
Keywords: AC220; Acute Myeloid Leukemia (AML); De Novo Acute Myeloid Leukemia (AML); Newly diagnosed Acute Myeloid Leukemia (AML); FMS-like tyrosine kinase (FLT3); FMS-like tyrosine kinase (FLT3) Inhibitor; Kinase; Kinase Inhibitor; Pharmacokinetics; ASP2689; quizartinib
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — quizartinib; Daunorubicin; Cytarabine; Cytosine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AC220 (Experimental)
  Interventions: Drug: AC220; Drug: daunorubicin; Drug: cytarabine

INTERVENTIONS:
Drug: AC220 — Oral Liquid
  Other Names: quizartinib; ASP2689
Drug: daunorubicin — Intravenous Infusion
  Other Names: Cerubidine; daunorubicin hydrochloride
Drug: cytarabine — Intravenous Infusion
  Other Names: Ara-C; Cytarabine Hydrochloride; Cytosar; Cytosine; Arabinoside

SUMMARY:
The purpose of this study is to define the maximum tolerated dose (MTD) of AC220 when combined with induction and consolidation therapy and as maintenance therapy following induction and consolidation.

DETAILED DESCRIPTION:
Subjects will receive escalating doses of AC220 plus standard 7+3 cytarabine and daunorubicin remission induction therapy. Subjects may receive up to 2 cycles of induction therapy. Subjects who have a complete response (including complete remission (CR) with incomplete hematologic recovery) are eligible to receive up to 3 consolidation cycles. In consolidation subjects will receive AC220 plus high dose cytarabine. Subjects achieving a composite Complete Remission (CRc) will be eligible to receive AC220 alone for up to 12 additional 28 day cycles.

Subjects will be enrolled into successive gender balanced cohorts of 6 subjects (at least 3 must be females) to determine the maximum tolerated dose (MTD). Dose escalation decision will be made based on dose limiting toxicities (DLTs) that occur during the first remission induction cycle. Seven and 14 day schedules will be evaluated.

After the MTD and schedule is established, the study will open to enroll between 14 to 34 subjects. Subjects will receive AC220 during induction and consolidation at the MTD and schedule established. Stopping rules will be used to evaluate safety at the current dose. If testing at a dose level must be stopped, then a lower dose may be tested. MTD will also be established for the maintenance therapy.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a diagnosis of previously-untreated de novo acute myeloid leukemia (AML) according to World Health Organization (WHO) classification (2008) documented within 28 days prior to enrollment and defined as > 20% myeloblasts on the marrow aspirate or peripheral blood differential, with or without extramedullary involvement, with confirmatory immunophenotyping or immunocytochemistry (e.g. myeloperoxidase). In addition, subjects with the clonal, recurring cytogenetic abnormalities: t(8;21)(q22;q22), inv(16)(p13q22) or t(16;16)(p13;q22) should be considered to have AML regardless of the blast percentage. Subjects with both positive and negative FMS-like tyrosine kinase - internal tandem duplication (FLT3-ITD) mutation status are eligible.
* Subject has an Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2.
* Subject must have adequate renal, hepatic, and coagulation parameters as indicated by the following laboratory values:
* Subject is a woman of childbearing potential (WOCBP) or a male subject with female partner of childbearing potential who agrees to use a medically-approved method of contraception to avoid pregnancy throughout the study and for at least 3 months after the last dose of study drug.
* Subject is a WOCBP and has a negative serum or urine pregnancy test (sensitivity ≤ 25 IU human chorionic gonadotropin [hCG]/L) within 72 hours prior to the start of study drug administration.
* Subject is able to comply with study procedures and follow-up examinations.

Exclusion Criteria:

* Subject has a diagnosis of acute promyelocytic leukemia (APL), French-American-British (FAB) classification M3 or World Health Organization (WHO) classification of APL with t(15;17)(q22;q12), or BCR-ABL positive leukemia (chronic myelogenous leukemia in blast crisis).
* Subject has a diagnosis of AML following an antecedent hematologic disorder (diagnosis of myelodysplasia or myeloproliferative neoplasm by bone marrow aspirate and/or biopsy documented at least 12 weeks prior to first dose of study drug).
* Subject has a diagnosis of acute bilineal/biphenotypic leukemia.
* Subject has therapy-related AML.
* Subject received previous treatment with AC220.
* Subject has received previous therapy for AML
* Subject has uncontrolled disseminated intravascular coagulation.
* Subject has Central Nervous System (CNS) leukemia. A Subject with symptoms suggestive of CNS leukemia must undergo a lumbar puncture; and subject with a positive cerebrospinal fluid (CSF) for AML blasts is not eligible.
* Subject has a known positive test for human immunodeficiency virus, hepatitis C, or hepatitis B surface antigen.
* Subject had major surgery within 4 weeks prior to the start of study drug.
* Subject has uncontrolled or significant cardiovascular disease - Subject has a pre-existing disorder predisposing the subject to a serious or life-threatening infection (e.g. cystic fibrosis, congenital or acquired immunodeficiency, bleeding disorder, or cytopenias).
* Subject has an active acute or chronic systemic fungal, bacterial, viral, or other infection.
* Subject has a concurrent disease (e.g. a history of serious organ dysfunction or disease) that may place the subject at undue risk to undergo induction therapy per protocol, or that might obscure assessments of drug safety.
* Subject requires treatment with concomitant drugs that prolong QT/QTc interval or strong cytochrome P-3A4 (CYP3A4) inhibitors or inducers with the exception of antibiotics, antifungals, and antivirals that are used as standard of care to prevent or treat infections and other such drugs that are considered absolutely essential for the care of the subject.
* Subject requires treatment with anticoagulant therapy.
* Subject is a female who is lactating.
* Subject has any medical, psychiatric, addictive or other kind of disorder which compromises the ability of the subject to give written informed consent and/or to comply with procedures.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2011-10; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Safety assessed by recording adverse events, physical examinations, vital signs, electrocardiograms (ECGs), and laboratory assessments | up to Day 42
Incidence of Dose Limiting Toxicity (DLT) | up to Day 42

SECONDARY OUTCOMES:
Pharmacokinetic assessment through analysis of blood samples | Up to Day 11

CONTACTS AND LOCATIONS:
Overall Officials: Guy Gammon, MB, BS, MRCP, Study Director — Medical Monitor, Ambit Biosciences Corporation
Locations (5):
- United States (5):
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - Northwestern University, Chicago, Illinois
  - Johns Hopkins Medical Institute, Baltimore, Maryland
  - Memorial-Sloan Kettering Cancer Center, New York, New York
  - M.D. Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/